CLINICAL TRIAL: NCT01772888
Title: Chewing Efficiency Measured by a Two Colour Chewing Gum Test: a Marker of Insufficient Nutritional Intakes and Percutaneous Gastrostomy (PEG) Necessity in ALS Patients?
Brief Title: Chewing Efficiency Measured by a Two Colour Chewing Gum Test in Amyotrophic Lateral Sclerosis (ALS) Patients?
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Genton Graf Laurence, MD, University Hospital, Geneva
Other Study IDs: 12-103
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis 11
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis 11

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with ALS: All subjects aged > 18 years, diagnosed with an ALS and included in the multidisciplinary follow-up of the HUG at time of diagnosis will be considered and included, if possible, at their first visit.
- Healthy age and gender-matched subjects: Controls matched for age and gender and dental status and without a medical history for neurological or otolaryngologic disease (1 control for 1 patient). They will be recruited among hospital staff and patients of the dental school.

SUMMARY:
Study aims: The primary aim is to determine whether chewing efficiency, determined by a two-colour mixing ability test, and maximum bite and lip force decrease in ALS patients.

DETAILED DESCRIPTION:
Study center: University Hospitals of Geneva Study type: Cohort study with matched controls Study population: 25 ALS patients included in the multidisciplinary cohort study of the University Hospital Geneva between October 2012 and October 2014 and followed for 3 years maximum and 25 controls, matched for age, sex and dental status.

Study duration: Inclusion from October 2012 to October 2016. Follow-up for 3 years.

Study hypothesis: Chewing efficiency, maximum bite and lip force decrease with time in ALS patients and may be a marker of texture adaptation and PEG necessity.

Study aims: The primary aim is to determine whether chewing efficiency, determined by a two-colour mixing ability test, and maximum bite and lip force decrease in ALS patients.

The secondary aims are to determine, in ALS patients, whether:

* Maximum bite and lip force decrease.
* Chewing efficiency, maximum bite and lip force decrease more in ALS patients with bulbar than with spinal onset.
* Chewing efficiency and bite force correlate with energy intakes, nasofibroscopic assessment, and a validated swallowing questionnaire.
* Saliva volume increases with time and progression of disease and influences masticatory efficiency.
* Saliva volume is associated with nasofibroscopy assessment.

Methods : Every three months, we will perform:

* As part of the ongoing cohort study (already accepted by the Ethical Committee) calculation of energy intakes through a 24h recall, nasofibroscopy, swallowing questionnaire and score of disease severity.
* As part of this study: assessment of dental status at first visit, chewing efficiency test by a with a colour mixing ability test, maximum voluntary bite and lip force, saliva volume and calculation of a 3-day dietary recall instead of a 24h recall.

Statistics: Evolutions with time and between groups, of chewing efficiency, bite and lip force will be assessed by repeated measures ANOVA. Correlations between two continuous variables will be examined by Spearman's correlation coefficients at the different time points. Correlations between a continuous variable and a binary variable (nasofibroscopic assessment) will be explored by logistic regression with mixed effect model.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients
* > 18 years
* Participation in the cohort study

Exclusion Criteria:

* Refusal of participating in the cohort study
* Presence of PEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS patients participating in the cohort study of the University Hospital Geneva
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
- Chewing efficiency | 5 years

SECONDARY OUTCOMES:
Lip force | 5 years
Bite force | 5 years
Calorie and protein intakes | 5 years
Saliva volume | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Schimmel M, Christou P, Herrmann F, Muller F. A two-colour chewing gum test for masticatory efficiency: development of different assessment methods. J Oral Rehabil. 2007 Sep;34(9):671-8. doi: 10.1111/j.1365-2842.2007.01773.x. PMID 17716266
- [Derived] Schimmel M, Leuchter I, Heritier Barras AC, Leles CR, Abou-Ayash S, Viatte V, Esteve F, Janssens JP, Mueller F, Genton L. Oral function in amyotrophic lateral sclerosis patients: A matched case-control study. Clin Nutr. 2021 Aug;40(8):4904-4911. doi: 10.1016/j.clnu.2021.06.022. Epub 2021 Jun 28. PMID 34358835